CLINICAL TRIAL: NCT03975738
Title: Map Healthcare Provision Outside the NHS Through the Development of Virtual Online Practice Communities in Primary and Secondary Care (VOICE)
Brief Title: Map Healthcare Provision Outside the NHS
Acronym: VOICE
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019SUR106
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Healthcare Providers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- A GP Surgery: A selection of healthcare workers from a GP Surgery to be recruited
  Interventions: Other: To be part of a blog
- A Patient and Public Involvement and Engagement Group: A selection of healthcare workers from a Patient and Public Involvement and Engagement Group to be recruited
  Interventions: Other: To be part of a blog
- Young Person's Steering Group: A selection of patients from a Young Person's Steering Group to be recruited
  Interventions: Other: To be part of a blog
- An Acute Trust: A selection of healthcare workers from an Acute Trust to be recruited
  Interventions: Other: To be part of a blog
- Hayward Hospital Social Care Team: A selection of healthcare workers from the Hayward Hospital Social Care Team to be recruited
  Interventions: Other: To be part of a blog
- A Hospice: A selection of healthcare workers from a Hospice to be recruited
  Interventions: Other: To be part of a blog
- West Midlands Cares: A selection of healthcare workers from a the West Midlands Cares Group to be recruited
  Interventions: Other: To be part of a blog
- CRN Clinical Research Speciality Leads (CRSL): A selection of healthcare workers from a group of CRN (Clinical Research Network) Clinical Research Speciality Leads (CRSL) to be recruited
  Interventions: Other: To be part of a blog
- CRN Sub Speciality Leads (SSL): A selection of healthcare workers from a CRN Sub Speciality Leads (SSL) to be recruited
  Interventions: Other: To be part of a blog
- A District General Hospital: A selection of healthcare workers from a A District General Hospital to be recruited
  Interventions: Other: To be part of a blog

INTERVENTIONS:
Other: To be part of a blog — To be part of a blog - to respond to questions and free to comment on other participants comments

SUMMARY:
* To collect data to show which sites outside of the NHS are currently being signposted to patients by Healthcare Multidisciplinary Professionals
* To collect data about these sites, from patients who have been referred or signposted to sites outside of the NHS from a Healthcare Multidisciplinary Professional
* To develop a database of potential healthcare sites outside the NHS that could become involved in NIHR Healthcare

DETAILED DESCRIPTION:
This is a small-scale pilot project to test out the research design and methodology. This pilot project will take a small-scale approach to mapping non-NHS providers that are currently (a) being recommended and signposted by healthcare professionals and (b) have been experienced by patients. A sample of around 100 participants who are (a) currently employed in a range of healthcare provision settings or who (b) have experienced healthcare provision outside the NHS and who (i) have regular access to internet access in order to access a blog; and (ii) have sufficient English language skills to read and understand questions posted on the blog, will be recruited.

Participants will be asked to provide information via a blog about which non-NHS healthcare provision they would signpost or recommend. There will be opportunities both to record data and to communicate and form discussions with other participants on the blog. This data will be coded and collated onto a database and analysed thematically.

ELIGIBILITY:
Inclusion Criteria:

* currently employed in a healthcare setting in a role that involves direct contact with patients for at least one day per week or
* have been a patient accessing non-NHS healthcare provision within the last two years.
* must have self-reported, sufficient English language ability to read the blog
* have regular personal access to the internet.

Exclusion criteria:

* not currently employed in a healthcare setting in a role that involves direct contact with patients for at least one day per week or
* not have been a patient accessing non-NHS healthcare provision within the last two years.
* not have self-reported, sufficient English language ability to read the blog
* not have regular personal access to the internet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participant Groups will be selected according to geographical location (within the West Midlands)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of health care practice in non-NHS sites | 5 months
  Questionnaire via a blog

CONTACTS AND LOCATIONS:
Overall Officials: Marion Evans, Principal Investigator — National Institute for Health Research, United Kingdom
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data to be shared with other researchers